CLINICAL TRIAL: NCT05374915
Title: An Open-Labeled, Single Arm Phase 2 Efficacy and Safety Study of REM-001 Photodynamic Therapy (PDT) for Treatment of Cutaneous Metastatic Breast Cancer (CMBC) That is Refractory or Not Eligible for Radiotherapy or Surgery
Brief Title: Efficacy and Safety Study of REM-001 Photodynamic Therapy for Treatment of Cutaneous Metastatic Breast Cancer (CMBC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kintara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTI-21-01
Record Dates: First submitted 2022-05-09; First posted 2022-05-16 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-11

CONDITIONS: Cutaneous Breast Cancer
Keywords: metastatic; cutaneous
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- REM-001 photodynamic therapy (PDT) (Experimental): Single arm study. All enrolled patients receive REM-001 therapy
  Interventions: Combination Product: REM-001 photodynamic therapy

INTERVENTIONS:
Combination Product: REM-001 photodynamic therapy — Infusion of REM-001 (iv) followed by light treatment to treatment field 24 hrs after infusion of REM-001

SUMMARY:
This is an open-label, single cohort study to confirm dose, assessments and timing of response, to support future studies. The primary objective of the trial is to evaluate cutaneous tumor response within total target treatment field to REM-001 therapy assessed using standardized digital photography

DETAILED DESCRIPTION:
All participants must have stable or responding systemic disease for at least 3 months at screening.

REM-001 Therapy:

Day 1: REM-001 = 0.8 mg/kg (IV) at 2 mL/Kg/hr (over approximately 24 minutes)

Day 2: Light treatment per treatment area= 100 J/cm2 (10 min per treatment field) - 24 hrs (± 2 hrs) after infusion of REM-001.

Total area of target lesions treated will be < 200 cm2. Participants will be assessed at week 1, 4, 8, 12, 16, 20 and 24 weeks. An additional 4 weeks follow up will be undertaken if confirmatory assessment is required after week 24.

Assessments will include:

* cutaneous lesion response using photographic imaging
* area of ulceration using photographic imaging
* presence or absence of ulceration, bleeding, discharge and eschar
* patient-reported assessments for pain and itch, using numeric rating scales
* quality of life assessments
* safety On Day 1 of treatment, the participant will undergo an ECG assessment post-infusion and a blood sample for determination of concentration of REM-001 in plasma will be collected post-infusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 18 years of age or greater.
* Participants able and willing to sign informed consent.
* Histopathologically confirmed breast cancer metastasis to the skin.
* Cutaneous metastasis not suitable for surgical resection.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Symptomatic lesions (including discomfort, pain, discharge, ulceration).
* Cutaneous, subcutaneous soft tissue, or superficial lymphatic metastasis that is amenable to PDT:

  * Lesion(s) > 10 mm and < 60 mm in longest dimension.
  * Lesion(s) exhibit at least one of the following symptoms: ulcerated, bleeding, discharging, itchy, painful.
  * Judged by investigator as eligible for PDT.
* Participants are radiotherapy refractory (have received a radiation dose of 60 gray (Gy) or greater to the ipsilateral thorax) or are not otherwise amenable to radiotherapy.
* Disease progression on at least 2 courses of systemic therapy:

  * HR positive/HER2 negative participants: should be refractory to endocrine therapy (at least 2 different regimens including at least one CDK4/6 inhibitor). Maintenance endocrine therapy at the clinician's discretion is allowed.
  * HER2 positive participants should have had disease progression on at least 2 different regimens of HER2 targeted therapies. Maintenance therapy on trastuzumab (HERCEPTIN®) is allowed.
* If participants are on systemic therapy at enrollment, they must meet the following:

  * Participants must have undergone a minimum of two cycles of systemic therapy prior to enrollment.
  * The systemic therapy must be one from the Treatment of Physician's Choice (TPC) list, as follows: : eribulin mesylate (Halaven®); capecitabine (Xeloda®); Gemcitabine (Gemzar®); a taxane [either docetaxel (Taxotere®), nab-paclitaxel (Abraxane®), or paclitaxel (Taxol®)]; vinorelbine (Navelbine®); an antibody-drug conjugate [either sacituzumab-govitecan (Trodelvy®), trastuzumab-deruxtecan (Enhertu®), or ado-trastuzumab emtansine (KADCYLA®)]; pembrolizumab (Keytruda®); or carboplatin (Paraplatin®).
  * Patients who are not on any chemotherapy will also be eligible.
* At the time of enrolment, participants should have no known plans to change or modify their TPC regimen while receiving study treatment. Note: TPC regimen may be changed or modified after treatment with REM-001 therapy, but this should be done in consultation with the Sponsor Medical Monitor.
* Adequate renal function, as evidenced by estimated glomerular filtration rate (eGFR) > 45 mL/min/1.73 m2 using the CKD-EPI Creatinine Equation without race.
* Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, hemoglobin ≥ 8.5 g/dL and platelet count ≥ 100 × 10^9/L; INR < 1.5.
* Adequate liver function as evidenced by bilirubin ≤ 2.0 times the upper limits of normal (ULN) and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 3 × ULN (in the case of liver metastases ≤ 5 × ULN) [Participants with known Gilbert's Syndrome who have serum bilirubin < 1.5 x ULN (NCI CTCAE v5.0 Gr 2) may be enrolled].
* QTCF < 470msec on baseline ECG
* Woman of childbearing potential (WOCBP) must have a negative serum pregnancy test documented within 7 days prior to registration and must agree to practice adequate contraception
* Male patients must be sterile or willing to use an approved method of contraception from the time of treatment with REM-001 until 90 days after study drug treatment.

Exclusion Criteria:

* Participants who have received local cryotherapy, radiotherapy, intra-lesional chemotherapy, systemic or topical PDT, or surgery to study lesion fields within the past 12 weeks.
* Participants with progressive brain or subdural metastases, or leptomeningeal disease.
* Participants with previously treated brain or subdural metastases may participate provided:

  * Previously treated brain metastases are stable and without evidence of progression, as determined by contrast-enhanced CT or MRI brain scan, for at least 4 weeks prior to the first dose of study treatment.
  * There is no evidence of new brain metastases
  * They have completed local therapy and discontinued the use of corticosteroids for this indication for at least 4 weeks prior to first dose of study treatment.
  * Any neurologic symptoms attributed to brain metastases must have been stable for at least 4 weeks prior to study enrollment
* History of allergic or hypersensitivity reactions to light, egg proteins or egg yolk; history of porphyria, systemic lupus erythematosus, or xeroderma pigmentosum.
* Known disorder of lipoprotein metabolism or clearance (cholesterol> 400 mg/dl, and/or triglycerides > 500 mg/dl).
* Participants who have received investigational agents within the past 4 weeks or within 4 half-lives of the investigational agent (whichever is shorter) before the first study drug dose.
* Participants with inflammatory breast cancer.
* Known human immunodeficiency virus (HIV) infection with detectable virus titer.
* Active or chronic hepatitis B or C infection.
* Active or ongoing infection requiring systemic treatment.
* Participants who have undergone major surgery within 4 weeks of study treatment, or have planned surgery within 4 weeks of anticipated initiation of treatment with REM-001 therapy.
* Participants with otherwise unexplained weight loss (> 10% body weight) in the last 30 days prior to Screening.
* History of other malignancy treated with curative intent within the last 3-5 years. Exceptions are: Curatively treated basal cell/squamous cell skin cancer; carcinoma in situ of the cervix; superficial transitional cell bladder carcinoma
* Patients with other major or uncontrolled medical conditions, e.g., myocardial infarction or New York Heart Association (NYHA) Class III/IV heart failure within the last 6 months, stroke, uncontrolled diabetes, uncontrolled autoimmune disease.
* WOCBP that is pregnant or breast-feeding, or planning to become pregnant or breast-feed during protocol treatment and for 3 months after last dose of REM-001 therapy.
* WOCBP unwilling to use effective contraception during protocol treatment and for 3 months after last dose of REM-001 therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Best Overall Objective Response Rate (bORR) | Up to week 24
  Best Overall Objective Response Rate (bORR) [complete response (CR) or partial response (PR)] of target treatment fields at any time from treatment up to, and including, week 24.

SECONDARY OUTCOMES:
Duration of best overall objective response | Up to week 24
  Duration of best overall objective response (CR or PR) based on initial target fields
Time from baseline to the date of the first objective response (PR or CR) | Up to week 24
  Time from baseline to the date of the first objective response (PR or CR)
Change from baseline in area of ulceration | Up to week 24
  How much the area of ulceration of initial target fields changes from that measured at baseline, when measured by standardized and calibrated digital photography.
Change from baseline in area and volume of lesions | Up to week 24
  How much the area and volume of lesions of initial target fields changes from that measured at baseline when measured by the standardized and calibrated 3D digital photography
Change from baseline in lesion discharge | Up to week 24
  Presence or absence of discharge of cutaneous lesion in initial target treatment field - investigator and independent review of photographs.
Change from baseline in lesion bleeding | Up to week 24
  Presence or absence of bleeding of cutaneous lesion in initial target treatment field - investigator and independent review of photographs.
Change from baseline in lesion eschar | Up to week 24
  Presence or absence of eschar of cutaneous lesion in initial target treatment field - investigator and independent review of photographs.
Change from baseline in patient reported assessment of pain | Up to week 24
  Improvement or worsening of severity of pain using the Brief Pain Inventory-Short Form (BPI-SF) questionnaire over 24 weeks from start of treatment
Change from baseline in patient reported assessment of itch | Up to week 24
  Improvement or worsening of severity of itching using the Pruritus numerical rating scale (NRS) questionnaire over 24 weeks from start of treatment
Change from baseline participant-reported overall quality of life | Up to week 24
  Improvement or worsening over 24 weeks from start of treatment in participant-reported overall quality of life assessed using the EORTC QLQ-C30 (v3.0) questionnaire
Investigator-assessed objective response rate (ORR) | Up to week 24
  Investigator-assessed objective response rate (ORR) over of target treatment fields at any time from treatment up to and including week 24
Progression Free Survival (PFS) | Up to week 24
  Progression Free Survival (PFS) of systemic disease based on RECIST 1.1
Overall Survival (OS). | Up to week 24
  Overall Survival (OS).
Adverse events | Up to week 24
  Incidence and severity of adverse events using CTCAE v5.0 until 24 weeks from treatment
Safety assessments | Up to week 24
  Incidence and severity of clinically significant safety assessments: clinical laboratory examinations, vital signs, and physical exam
Electrocardiogram (ECG) - QT interval | Day 1 and 2
  The effect of REM-001 therapy on QT interval post-infusion
Plasma concentrations of REM-001 | Day 1 and 2
  Determination of plasma concentrations of REM-001 at the end of infusion (15 min post-infusion on day 1) and 24 hrs post-infusion prior to light treatment on day 2

CONTACTS AND LOCATIONS:
Overall Officials: Alina Markova, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No